CLINICAL TRIAL: NCT01027390
Title: Work Place Adjusted Intelligent Physical Exercise Reducing Musculoskeletal Pain in Shoulder and Neck (VIMS, Danish Acronym)
Brief Title: Work Place Adjusted Intelligent Physical Exercise Reducing Musculoskeletal Pain in Shoulder and Neck
Acronym: VIMS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: National Research Centre for the Working Environment, Denmark (Other Government); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Gisela Sjogaard, Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-C-2008-103; NCT01056068 (obsolete NCT alias)
Record Dates: First submitted 2009-12-07; First posted 2009-12-08 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Musculoskeletal Disorders
Keywords: neck/shoulder
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 hr training 50% supervision (Experimental): 1 hr training 50% supervision
  Interventions: Behavioral: physical training exercise
- 3 x 20 min training 50% supervision (Experimental): 3 x 20 min training 50% supervision
  Interventions: Behavioral: physical training exercise
- 3 x 20 min training initial instructions (Experimental): 3 x 20 min training initial instructions
  Interventions: Behavioral: physical training exercise
- 10 x 6 min training 50% supervision (Experimental): 10 x 6 min training 50% supervision
  Interventions: Behavioral: physical training exercise
- reference (No Intervention): no training

INTERVENTIONS:
Behavioral: physical training exercise — physical exercise training at the work site during work time
  Arms: 1 hr training 50% supervision; 10 x 6 min training 50% supervision; 3 x 20 min training 50% supervision; 3 x 20 min training initial instructions

SUMMARY:
Musculoskeletal disorders are frequent among office workers especially in the neck/shoulder area.

The hypothesis is, that specific strength training of the neck/shoulder muscles will alleviate the pain.

The two sub-hypotheses are

1. Alleviation of pain is independent of training frequency
2. Alleviation of pain is higher following supervised training vs training with initial instruction only

DETAILED DESCRIPTION:
Recent studies have shown a positive effect of work site physical exercise intervention, however, there is a lack of evidence regarding: 1) extend of instruction and supervision, and 2) frequency of training session during the wek.

Questionnaires will be send to around 2000 office workers inviting them to participate in work site training for 1 hr per week for 20 weeks. Those accepting the invitation will be randomized into 5 different groups:

1. training 1 hr one time per week supervized 50% of the time
2. training 3 x 20 min per week supervised 50 % of the time
3. training 3 x 20 min per week supervised only initially with careful instructions
4. training 10 x 6 min per week supervised 50 % of the time
5. no training serving as reference control group At termination of the training period there will be a follow-up questionnaire survey

ELIGIBILITY:
Inclusion Criteria:

* office workers
* employed

Exclusion Criteria:

* physically heavy work
* trauma
* leif threatening disease, e.g. cancer,
* pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 573 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
neck/shoulder pain, selfreported | 20 weeks

SECONDARY OUTCOMES:
muscle strength and endurance | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gisela Sjogaard, Dr.Med.Sci., Principal Investigator — University of Southern Denmark
Locations (1):
- Rigspolitiet, Copenhagen, Denmark

REFERENCES:
- [Result] Andersen CH, Andersen LL, Gram B, Pedersen MT, Mortensen OS, Zebis MK, Sjogaard G. Influence of frequency and duration of strength training for effective management of neck and shoulder pain: a randomised controlled trial. Br J Sports Med. 2012 Nov;46(14):1004-10. doi: 10.1136/bjsports-2011-090813. Epub 2012 Jun 29. PMID 22753863
- [Result] Andersen LL, Zebis MK, Pedersen MT, Roessler KK, Andersen CH, Pedersen MM, Feveile H, Mortensen OS, Sjogaard G. Protocol for work place adjusted intelligent physical exercise reducing musculoskeletal pain in shoulder and neck (VIMS): a cluster randomized controlled trial. BMC Musculoskelet Disord. 2010 Aug 5;11:173. doi: 10.1186/1471-2474-11-173. PMID 20687940
- [Derived] Dalager T, Bredahl TG, Pedersen MT, Boyle E, Andersen LL, Sjogaard G. Does training frequency and supervision affect compliance, performance and muscular health? A cluster randomized controlled trial. Man Ther. 2015 Oct;20(5):657-65. doi: 10.1016/j.math.2015.01.016. Epub 2015 Feb 28. PMID 25816746